CLINICAL TRIAL: NCT00661089
Title: "A Randomized Double-Blind Placebo-Controlled Trial of Botulinum Toxin Type A (BOTOX ) in the Treatment of Hemiplegic Shoulder Pain and Spasticity"
Brief Title: Randomized DB Controlled Trial of Botulinum Toxin A in Hemiplegic Shoulder Pain and Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Christina Marciniak, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0335-006
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2012-02-06 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Post-stroke Shoulder Pain and Spasticity
Keywords: stroke; shoulder pain; spasticity
MeSH Terms: conditions — Muscle Spasticity; Stroke; Shoulder Pain | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular OnabotulinumtoxinA (Experimental): Injection of Botulinum Toxin type A - onabotulinumtoxinA into specified shoulder muscles at second visit
  Interventions: Drug: Botulinum Toxin Type A - OnabotulinumtoxinA
- Intramuscular Placebo (Saline) (Active Comparator): Injection of saline into specified shoulder muscles at Visit 2. Blind broken and subjects were offered study drug if initially in the placebo group, at week 12
  Interventions: Drug: Placebo (Saline)

INTERVENTIONS:
Drug: Botulinum Toxin Type A - OnabotulinumtoxinA — 100-200 units injected into the pectoralis major. The teres major may also be injected if tone is noted in shoulder extensors.
  Other Names: BOTOX
  Arms: Intramuscular OnabotulinumtoxinA
Drug: Placebo (Saline) — Equivalent volume of saline without study drug injected into the pectoralis major. Teres major was also injected if tone noted in the shoulder extensors.
  Arms: Intramuscular Placebo (Saline)

SUMMARY:
The purpose of this study is to evaluate whether botulinum toxin type A injected into muscles around the shoulder is effective in treating shoulder pain and improving function in patients with shoulder pain and involuntary muscle tightness after a stroke.

DETAILED DESCRIPTION:
Subjects with shoulder pain and spasticity at the shoulder following a stroke resulting in hemiplegia are eligible for participation. Following an initial screening visit involving a history and physical examination, subjects will be entered in to the study if they have significant spasticity of shoulder internal rotation/adduction associated with pain rated at least a 4 on the VAS for pain. Subjects will also be given a cognitive screening in which they will be asked to rate pain in hypothetical situations.

Shoulder pain is a frequent complication following hemiplegic stroke, and may result in further disability. Spasticity is also a complication following stroke . Botulinum toxin is used in the treatment of post-stroke spasticity and may also have pain modulating effects. Participants in this study will be asked to make total of 6 visits over a period of approximately 13 weeks. Eligible subjects will be randomized to 100 to 200 units of botulinum toxin type injected into the pectoralis major at the second visit. If there is significant spasticity for shoulder extension, subjects will also receive injections into the teres major. Subjects will be followed up with assessments of pain, functioning, active and passive range of motion and depression following the initial injection. At the 12 weeks post injection visit, the blinding will be broken and subjects initially injected with placebo will be injected with the active drug. This will be done to give all subjects an opportunity to receive the active drug, as well as to assess the effects of any differences with delayed treatment. All subjects will return 4 weeks later to repeat the same assessments above. Subjects will be called at one year post study enrollment for repeat pain ratings and for information regarding subsequent treatments.

.

ELIGIBILITY:
Inclusion Criteria:

* Post stroke greater than 2 months
* Shoulder pain despite PT/OT interventions
* Weight greater than 88 lbs
* Stable medically
* Spasticity

Exclusion Criteria:

* Myasthenia gravis or other medical conditions that preclude use of botulinum toxin
* Pregnancy
* Infection or dermatologic conditions at the injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-09; Primary Completion 2009-03 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Marciniak, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Marciniak CM, Harvey RL, Gagnon CM, Duraski SA, Denby FA, McCarty S, Bravi LA, Polo KM, Fierstein KM. Does botulinum toxin type A decrease pain and lessen disability in hemiplegic survivors of stroke with shoulder pain and spasticity?: a randomized, double-blind, placebo-controlled trial. Am J Phys Med Rehabil. 2012 Dec;91(12):1007-19. doi: 10.1097/PHM.0b013e31826ecb02. PMID 23064478

RESULTS

PARTICIPANT FLOW:
Groups:
- onabotulinumtoxinA Injection: Botulinum Toxin injected at second visit
- Saline Injection: Receives placebo injections following randomization (Saline).Delayed treatment group.
  Blind broken and receives botulinum toxin at week 12
Period: Overall Study
Arm/Group | onabotulinumtoxinA Injection | Saline Injection
Started | 10 | 11
Completed | 10 | 9
Not Completed | 0 | 2
Not completed — 1 subject withdrawal | 0 | 1
Not completed — death at 8 weeks due to new stroke | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA Injection | Saline Injection | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.8) | 58.9 (10.3) | 60.00 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Secondary Outcome: Change in Disability Assessment Scale for Hygiene
Description: Subject rating of scores on the Disability Assessment Scale Range 0-3, Minimum value 0= no disability, Maximum value 3= severe disability Higher Score indicates worse outcome
Time Frame: baseline and 4 weeks post injection
Population: All enrolled subjects completed the baseline and for week post-injection measurements for this outcome
Measure: Median (Inter-Quartile Range); unit: Score on a scale from 0-3
Groups:
- Placebo: Group recieved saline injections intramuscularly of equivalent volume
- Botulinum Toxin Injection: Group received botulinum toxin type A (Botox) in the pectoralis and teres major muscles
Arm/Group | Placebo | Botulinum Toxin Injection
Number analyzed (Participants) | 11 | 10
Score on a scale from 0-3 | 1.0 [0 to 1.5] | -1.0 [-1.0 to 0]

2. Secondary Outcome: Time to Don a Pull Over Shirt
Time Frame: 2,4,12, and 16 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Ability to Perform Hygiene Rating
Time Frame: 2,4,12, and 16 weeks
Reporting Status: Not Posted

4. Primary Outcome: Change in Pain Rating From Baseline to Four Weeks
Description: Change scores from patient ratings on the Visual Analogue Scale on 101 mm scale for worst pain, averaged over a week. Ratings performed at baseline and week four. Scale range 0-100 mm. Minimum value 0= No pain, Maximum value 100= worst pain Higher score indicates worse outcome
Time Frame: baseline and four weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Placebo: Group received saline injections intramuscularly of equivalent volume
Arm/Group | Placebo | Botulinum Toxin Injection
Number analyzed (Participants) | 11 | 10
units on a scale | -19.88 [-69.90 to 2.16] | -18.64 [-29.73 to 2.14]

ADVERSE EVENTS:
Time Frame: From enrollment through 12 weeks post injection
Arm/Group | onabotulinumtoxinA Injection | Saline Injection
Serious Adverse Events (participants affected / at risk) | 1/10 | 4/11
Other Adverse Events (participants affected / at risk) | 1/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | onabotulinumtoxinA Injection (N=10) | Saline Injection (N=11)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2) — Subjects were asked at each visit for any adverse effects. 1 subject with UTI requiring hospitalization
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Rectal bleeding requiring hospitalization
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Anemia requiring hospitalization and transfusion
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
New Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | onabotulinumtoxinA Injection (N=10) | Saline Injection (N=11)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2) — Urinary tract infection not requiring hospitalization
depression (Psychiatric disorders) | 1 (1) | 0 (0) — Depressive symptoms noted on Beck Depression, referred to psychology

LIMITATIONS AND CAVEATS:
Best and Worst pain collected, which may have limited the ability to detect overall pain. At the time of enrollment, subjects were on average very impaired by the Fugl-Meyer Scale measure, and pain on average had been present for several years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No